CLINICAL TRIAL: NCT02197494
Title: An Open Label, Balanced, Randomized, Two-treatment, Two Period, Two-sequence, Single Oral Dose, Crossover, Bioequivalence Study of Two Formulations of Valsartan 320mg Tablet in Healthy, Adult, Human Subjects Under Fed Condition.
Brief Title: Bioequivalence Study of Valsartan 320mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 042-14
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Valsartan Tablets USP 320 mg DIVIS
  Interventions: Drug: Valsartan
- Reference (Active Comparator): Diovan® (Valsartan) 320 Tablets
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan — 320mg tablets

SUMMARY:
The study was an open label, balanced, randomized, two-treatment, two-period, two sequence, single oral dose, crossover, bioequivalence study of two formulations of Valsartan 320 mg under fed conditions.

DETAILED DESCRIPTION:
After an overnight fast of at least 10 hours, the subjects were served a USFDA recommended high fat high calorie non-vegetarian breakfast, which they consumed within 30 minutes.

A single oral dose (320 mg) of either the test or the reference product was administered to the subjects at 30 ± 2 minutes minutes after serving the USFDA recommended high fat high calorie non-vegetarian breakfast. The IMP was administered in sitting posture with 240 mL of drinking water at ambient temperature. The IMP administration was as per the randomization schedule and under open-label condition.

A total of twenty-six (26) blood samples including pre-dose sample (duplicate), each of 02 mL, were collected from each subject except for the discontinued / withdrawn subjects to analyze the pharmacokinetic profile of the test as well as the reference drug.

The pharmacokinetic parameters were calculated from the drug concentration vs. time profile by non-compartmental model using WinNonlin Professional Software Version 5.3 (Pharsight Corporation, USA) for Valsartan. Statistical comparison of the pharmacokinetic parameters of the two formulations was carried out using PROC MIXED of SAS® Version 9.3 (SAS Institute Inc., USA) to assess the bioequivalence of both the formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, human volunteers between 18 to 45 years of age (both inclusive) living in and around Mumbai city or western part of India.
2. Having a Body Mass Index (BMI) between 18.5 - 24.9 (both inclusive), calculated as weight in kg/height in meter2.
3. Not having any significant disease in medical history or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12- lead ECG and X-ray chest (P/A view) recordings.
4. Able to understand and comply with the study procedures, in the opinion of the investigator.
5. Able to give voluntary written informed consent for participation in the trial.
6. In case of female subjects:

   * Surgically sterilized at least 6 months prior to study participation; Or
   * If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.

And

• Pregnancy test must be negative.

Exclusion Criteria:

1. Known hypersensitivity or idiosyncratic reaction to valsartan or any of the formulation excipients or any related drug.
2. History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
3. Sitting blood pressure less than 110 /70 mm Hg and pulse rate less than 60 or more than 100 beats per minute at the time of screening.
4. Presence of orthostatic hypotension.
5. If the QTc interval were to be more than 450 ms on ECG measurement at the time of screening.
6. Ingestion of a medicine (including herbal remedies) at any time within 14 days before dosing in period-I. In any such case subject selection were at the discretion of the Principal Investigator.
7. Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
8. A recent history of harmful use of alcohol (less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to receiving study medicine.
9. Smokers, who smoke 10 or more than 10 cigarettes/day or inability to abstain from smoking during the study.
10. The presence of clinically significant abnormal laboratory values during screening.
11. Use of any recreational drugs or history of drug addiction or testing positive in pre study drug scans.
12. History or presence of psychiatric disorders.
13. A history of difficulty in donating blood.
14. Donation of blood (1 unit or 350 mL) or receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study.

    Note: In case the blood loss is ≤ 200 mL; subject may be dosed 60 days after blood donation or last sample of the previous study.
15. A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.
16. A positive test result for HIV antibody.
17. An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medicine in period-I. In any such case subject selection were at the discretion of the Principal Investigator.
18. Consumption of grapefruit or grapefruit products within 48 hours prior to dosing.
19. Nursing mothers (females).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of Valsartan | 0-36 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Lambda Therapeutic Research Ltd., Navi Mumbai, Maharashtra, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm